CLINICAL TRIAL: NCT03987373
Title: Compare the Efficacy of Different Antiplatelet Therapy Strategy After Coronary Artery Bypass Graft Surgery: Follow-up Extension
Brief Title: DACAB Trial: Follow-up Extension
Acronym: DACAB-FE
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Qiang Zhao,MD, Professor and director, Department of Cardiac Surgery,Vice President of Ruijin Hospital, Ruijin Hospital
Other Study IDs: ESR-18-13658
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Bypass Grafting; Antiplatelet Therapy
Keywords: CABG; Antiplatelet; MACE; grafts patency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non-interventional — This study is a non-interventional, observational study. After completing 12-month treatment from DACAB trial, investigators would not make any interventions or impact on subjects' therapeutic strategy.

SUMMARY:
This study will include the subjects who enrolled in DACAB trial (NCT02201771) to observe clinical outcomes 5 years after coronary artery bypass grafting（CABG）.

The primary objective is to compare the occurrence of MACE-4 ( a composite of all-cause death, myocardial infarction, stroke, and coronary revascularization) among 3 randomized regimens (T+A, T alone, A alone) in previous DACAB trial within 5 years after CABG.

The secondary objectives are to compare the occurrence of MACE-5( a composite of all-cause death, myocardial infarction, stroke, coronary revascularization and hospitalization for unstable angina); MACE-3 ( a composite of cardiovascular death, myocardial infarction, and stroke); all-cause death; cardiovascular death; myocardial infarction; stroke; coronary revascularization; hospitalization for unstable angina and grafts patency rate among 3 randomized regimens in previous DACAB trial within 5 years after CABG.

The exploratory objectives are to compare the occurrence of MACE-4; MACE-5; MACE-3; all-cause death; cardiovascular death; myocardial infarction; stroke; coronary revascularization and hospitalization for unstable angina between 2 cohorts with or without grafts/vein grafts failure at 1 year angiographic follow-up.

DETAILED DESCRIPTION:
This is a non-interventional, observational study designed to compare clinical outcomes 5 years after CABG in subjects enrolled in DACAB trial.

After completing 12-month randomized treatment from DACAB trial, investigators would not make any interventions or impact on subjects'therapeutic strategy. Aspirin monotherapy would be given to most subjects according to the current guidelines. However, other antiplatelet regimens might be given for subjects by their attending physician based on the subject's individual condition. Subjects would spontaneously undergo regular laboratory test , electrocardiogram (ECG), ultrasound cardiography (UCG), coronary computed tomographic angiography (CCTA) or coronary angiography (CAG) and clinical follow-up according to clinical need and their individual condition. At 5-year (± 3 month) after CABG, a face-to-face visit is scheduled to be performed to collect the occurrence of clinical events, including types and time of events.

Some prospective exploratory analysis are planned. According to the 1-year angiographic outcome of all grafts from the DACAB trial, all subjects will be allocated to 2 non-randomized cohorts: Cohort A with at least one graft failure (Fitzgibbon Grade B or O) at 1 year, and Cohort B without any graft failure at 1 year. Then prospective exploratory analysis will be performed to compare the occurrence of MACE-4; MACE-5; MACE-3; and other outcomes between 2 non-randomized cohorts from 1-year angiographic follow-up to 5 years after CABG. Similar analysis will be performed according to the 1-year angiographic outcome of vein grafts only.

Other preplanned subgroup analysis included: baseline gender, baseline age stratification(70 years), baseline status of acute coronary syndrome, history of hypertension, baseline history of diabetes, baseline history of high-density lipoprotein cholesterol, baseline history of high-density lipoprotein (a) cholesterol, baseline history of prior myocardial infarction, baseline history of stroke, baseline history of peripheral vascular disease, Baseline history of COPD , baseline history of CKD-3 or above , baseline history of smoking, baseline left main coronary artery disease, baseline SYNTAX score stratification, baseline EuroSCORE stratification, baseline CABG with or without cardiopulmonary bypass, baseline CABG with or without internal thoracic artery grafts, baseline CABG with or without complete revascularization.

ELIGIBILITY:
Inclusion Criteria:

* This study will include the subjects who enrolled in DACAB trial

Exclusion Criteria:

* This study will include the subjects who enrolled in DACAB trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include the subjects who enrolled in DACAB trial
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
The time to the first MACE-4 event | within 5 year after CABG
  The time to the first occurrence of any MACE-4 event, defined as a composite of all-cause death, myocardial infarction, stroke and coronary revascularization.

SECONDARY OUTCOMES:
The time to the first MACE-5 event | within 5 year after CABG
  The time to first occurrence of any MACE-5 event, defined as a composite of all-cause death, myocardial infarction, stroke, coronary revascularization and hospitalization for unstable angina.
The time to the first MACE-3 event | within 5 year after CABG
  The time to first occurrence of any MACE-3 event, defined as a composite of cardiovascular death, myocardial infarction, and stroke.
The time to the first occurrence of all-cause death. | within 5 year after CABG
  The time to occurrence of any death
The time to the first cardiovascular death | within 5 year after CABG
  The time to occurrence of any cardiovascular death
The time to the first myocardial infarction | within 5 year after CABG
  The time to occurrence of any myocardial infarction, including STEMI, NSTEMI, or silent MI.
The time to the first stroke | within 5 year after CABG
  The time to occurrence of any stroke, including ischemic, hemorrhagic, or unknown type.
The time to the first coronary revascularization | within 5 year after CABG
  The time to occurrence of any repeated coronary revascularization, including PCI or CABG, no matter ischemic driven or not.
The time to the first hospitalization for unstable angina. | within 5 year after CABG
  The time to occurrence of any hospitalization for unstable angina. By definition, UA is cardiac biomarker negative with no evidence of AMI.
The rate of grafts failure (Fitzgibbon Grade B+O). | at 5 years after CABG ( if not available, at anytime within 5 year after CABG)
  assessed by CCTA or CAG, including artery and vein grafts.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Zhao, MD, Principal Investigator — Ruijin Hospital; Mario FL Gaudino, MD, Principal Investigator — Weill Cornell Medicine NewYork Presbyterian Hospital; Yunpeng Zhu, MD, Study Director — Ruijin Hospital
Locations (6):
- China (6):
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - Nan Jing First Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Xinhua Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhu Y, Zhang W, Dimagli A, Han L, Cheng Z, Mei J, Chen X, Wang X, Zhou Y, Xue Q, Hu J, Tang M, Wang R, Song Y, Kang L, Redfors B, Gaudino M, Zhao Q. Antiplatelet therapy after coronary artery bypass surgery: five year follow-up of randomised DACAB trial. BMJ. 2024 Jun 11;385:e075707. doi: 10.1136/bmj-2023-075707. PMID 38862179

DOCUMENTS (2):
  • Study Protocol (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT03987373/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT03987373/SAP_001.pdf